CLINICAL TRIAL: NCT00994487
Title: Breastfeeding, Parental Feeding Style, and Self-regulation Capabilities in Female Preschool-age Children
Brief Title: Breastfeeding in Infancy and Food Intake in Preschool-Aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 7828B
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Childhood Obesity; Breastfeeding
Keywords: Childhood Obesity; Breastfeeding; Bottle Feeding; Dietary Intake; Preload; Compensation; Parental Feeding Style
MeSH Terms: conditions — Pediatric Obesity; Breast Feeding; Bottle Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Breastfed child (Experimental): Female, normal weight, 3 to 5 year old children, exclusively breastfed from birth to 3 months of age
  Interventions: Other: High Energy Density Preload; Other: Low Energy Density Preload
- Bottle Fed Child (Active Comparator): Female, normal weight, 3 to 5 year old children, exclusively bottle fed from birth to 3 months of age
  Interventions: Other: High Energy Density Preload; Other: Low Energy Density Preload

INTERVENTIONS:
Other: High Energy Density Preload — Each child with a parent will attend a lunch session. In these sessions children will drink a liquid preload that is high in energy density and then they will consume an ad libitum lunch. The ad libitum lunch will be videotaped, and the videotapes will be coded for parental feeding styles
Other: Low Energy Density Preload — Each child with a parent will attend a lunch session. In these sessions children will drink a liquid preload that is low in energy density and then they will consume an ad libitum lunch. The ad libitum lunch will be videotaped, and the videotapes will be coded for parental feeding styles.

SUMMARY:
The purpose of this study is to compare female, preschool-aged children breastfed during infancy to female, preschool-aged children bottle-fed during infancy in their ability to adjust calorie intake in response to internal signals of hunger and fullness. Children and a parent will come to two sessions, with the children given drinks that are either high or low in energy, and then consume a lunch following the drink. The parent will be present during the lunch. Greater ability to self-regulate intake is demonstrated when less energy is consumed at lunch following the high energy drink as compared to the lunch following the low energy drink. Lunches will be videotaped so that parental feeding styles (i.e., how the parent interacted with the child during lunch) can be examined. The primary hypotheses are: 1.) the exclusively breastfed children will have higher self-regulation ability than the exclusively bottle-fed children, and 2.) the mothers of the exclusively breastfed children will demonstrate a parental feeding style characterized by less control and restriction than the mothers (or parent primarily responsible for child feeding) of the exclusively bottle-fed children.

DETAILED DESCRIPTION:
Research reports that children who were breastfed as infants have a decreased risk of becoming obese. However, it is not clear how breastfeeding may prevent the development of obesity. Breastfeeding may support the maintenance of sensitivity to internal hunger/fullness cues, which helps with self-regulating energy intake. Additionally, breastfeeding may facilitate the development of a parental feeding style low in control or restriction. This type of feeding style is also associated with greater ability to self-regulate energy intake. Bottle-feeding shifts feeding control to parents, and may lead to a parental feeding style high in control or restriction, impairing children's self-regulation abilities.

The aims of this study are to determine in females aged 3-5 years if: 1.) breastfed children have greater energy self- regulation capabilities; 2.) parents of breastfed children demonstrate a parental feeding style characterized by less control or restriction; and 3.) children with the greatest energy self-regulation capabilities were breastfed and have parents with feeding styles lowest in control or restriction. It is hypothesized that female, preschool-aged children breastfed and/or parented with a feeding style low in control or restriction self-regulate intake better than females not breastfed and/or parented with a feeding style high in control or restriction.

A within-subjects, counterbalanced design, using a standard preloading paradigm, will measure children's ability to self-regulate intake to preloads of differing energy densities. Children and a parent will participate in two trials, with children consuming preloads high and low in energy followed by a lunch in which energy intake is measured. Lunch will be videotaped so parental feeding style during the child's lunch can be coded for restriction and control. Results will provide information about potential mechanisms by which breastfeeding reduces the risk of obesity and obesity related diseases in children.

ELIGIBILITY:
Inclusion Criteria:

Children will be eligible for study participation if they meet the following criteria:

* female
* BMI between the 5th and the 85th percentile
* were of normal birth weight (>2500 g)
* full-term
* have no chronic disease conditions effecting growth and intake
* have not been in foster care for longer than one month (if at all)
* are between 3 and 5 years of age
* are willing to consume and are not allergic to the preloads and meals used in the study
* are not lactose-intolerant
* have a parent who is able to recall mode of feeding in infancy and was either exclusively breast-fed from birth to 3 months of age (defined as being fed from a bottle on average < 1 time per week from birth to 3 months of age, with all other feedings from the breast) or was exclusively bottle-fed from birth to 3 months of age (defined as being completely bottle-fed, with feedings comprised of formula and/or breastmilk)
* have a parent willing to transport child to the University of Tennessee lab at two different times during their participation in the project

Ages: 3 Years to 5 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Compensation for high energy density and low energy density preloads | 2 days

SECONDARY OUTCOMES:
Parental feeding style | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, Principal Investigator — University of Tennessee; Katie Kavanagh, PhD, Study Chair — Univerisity of Tennessee; Hiliary Fouts, PhD, Study Chair — University of Tennessee
Locations (1):
- University of Tennessee, Knoxville, Tennessee, United States

REFERENCES:
- See also: Website for the Healthy Eating and Activity Laboratory (HEAL) where the study is conducted — http://heal.utk.edu